CLINICAL TRIAL: NCT05631197
Title: Biomimetic Hydroxyapatite vs Fluoride for the Domiciliary Oral Hygiene of Pediatric Patients With Asthma and/or Allergic Rhinitis: Randomized Clinical Trial
Brief Title: Biomimetic Hydroxyapatite in Pediatric Patients With Asthma and/or Allergic Rhinitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-PEDOBIOREPAIR
Record Dates: First submitted 2022-11-18; First posted 2022-11-30 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Dental Caries; Periodontal Diseases
Keywords: Dental hygiene
MeSH Terms: conditions — Dental Caries; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Experimental)
  Interventions: Other: Biorepair Total Protection Plus + desensitizing enamel-repair shock treatment
- Control group (Active Comparator)
  Interventions: Other: Sensodyne Repair & Protect

INTERVENTIONS:
Other: Biorepair Total Protection Plus + desensitizing enamel-repair shock treatment — Domiciliary use twice a day
  Arms: Trial group
Other: Sensodyne Repair & Protect — Domiciliary use twice a day
  Arms: Control group

SUMMARY:
The aim of the study is to compare the incidence of dental caries and the level of demineralization in pediatric patients with asthma and/or allergic rhinitis.

Patients will conduct professional oral hygiene at the baseline. The following clinical indexes will be assessed: BEWE Index, Plaque Index, Bleeding Score, Schiff Air Index. Then, patients will be randomly divided into two groups:

* Trial group: domiciliary use of Biorepair Total Protection Plus + desensitizing enamel-repair shock treatment twice a day
* Control group: domiciliary use of Elmex Caries Protection twice a day

The clinical indexes will be assessed again after 1 month (T1), after 3 (T2) and 6 months (T3).

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients aged between 6-14 years
* diagnosis of allergic rhinitis and asthma
* therapy with salmeterol/fluticasone propionate
* diffused enamel demineralizations of deciduous and permanent teeth

Exclusion Criteria:

* low cooperation according to grades 3 and 4 of Frankl behavioral scale
* nonadherence to the study protocol checked by parents
* other systemic diseases.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Change of the BEWE Index - Basic Erosive Wear Examination (Barlet et al.2008) | Baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3)
  Scoring criteria:
  0 = no erosive tooth wear;
  1. = initial loss of surface texture;
  2. = distinct defect, hard tissue loss < 50% of the surface area;
  3. = hard tissue loss ≥ 50% of the surface area.
  The BEWE will be assessed with Intact Tooth application
Change in Shiff Air Index - Dental sensitivity test | Baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3)
  Scoring criteria:
  0 = the subject did not respond to air blasting;
  1. = the subject responded to air blasting;
  2. = the subject responded to air blasting and requested discontinuation;
  3. = the subject responded to air blasting, requested discontinuation and considered the stimulus to be painful.
Change in BoP - Bleeding on Probing | Baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3)
  Scoring criteria:
  Percentage of bleeding sites (mesial, distal, vestibular, lingual) of each teeth on the total available sites.
Change in PI - Plaque Index (Silness and Löe, 1964) | Baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3)
  Scoring criteria:
  0 = no plaque;
  1. = thin plaque layer at the gingival margin, only detectable by scraping with a probe;
  2. = moderate layer of plaque along the gingival margin; interdental spaces free, but plaque is visible to the naked eye;
  3. = abundant plaque along the gingival margin; interdental spaces filled with plaque.
Change in salivary pH | Baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3)
  Use of Just Fitter strips to assess salivary pH.
Change in SI - Susceptibility Index | Baseline (T0), 1 month (T1), 3 months (T2), 6 months (T3)
  Scoring criteria:
  * mild: 6.7< pH <7.8, BEWE 0-1, SAI 0-1
  * moderate: 6.0 <pH <6.6, BEWE 1-2, SAI 1-2
  * severe: pH <6.6, BEWE 2-3, SAI 2-3

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, MS, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.